CLINICAL TRIAL: NCT07129629
Title: Short-Course Regimen With Bedaquiline, Moxifloxacin and Pyrazinamide for Early Bactericidal Activity in Drug-Susceptible Tuberculosis
Acronym: Beams
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Huashan Hospital (Other); Guangzhou National Laboratory (Unknown)
Responsible Party: Principal Investigator, Wei Sha MD & PhD, Chief Physician and Doctoral Supervisor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beams Study
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis, Pulmonary; Drug-Susceptible Pulmonary Tuberculosis
Keywords: Bedaquiline; Moxifloxacin; Pyrazinamide; Early Bactericidal Activity; Drug-Susceptible Tuberculosis; Short-course regimen
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — bedaquiline; Moxifloxacin; Pyrazinamide; OPC-67683; Fumigant 93; Isoniazid; Protons; Rifampin; Ethambutol

STUDY DESIGN:
Masking Description: Not applicable - open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BZMD Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Delamanid) (Experimental): 4-month short-course regimen. Intensive phase (8 weeks): Bedaquiline + Pyrazinamide + Moxifloxacin + Delamanid. Consolidation phase (9 weeks): Bedaquiline + Moxifloxacin + Delamanid. Total treatment duration 17 weeks followed by follow-up until week 38.
  Interventions: Drug: Bedaquiline (B); Drug: Moxifloxacin; Drug: Pyrazinamide (PZA); Drug: Delamanid (D)
- BZMH Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Isoniazid) (Experimental): 4-month short-course regimen. Intensive phase (8 weeks): Bedaquiline + Pyrazinamide + Moxifloxacin + Isoniazid. Consolidation phase (9 weeks): Bedaquiline + Moxifloxacin + Isoniazid. Total treatment duration 17 weeks followed by follow-up until week 38.
  Interventions: Drug: Bedaquiline (B); Drug: Moxifloxacin; Drug: Pyrazinamide (PZA); Drug: Isoniazid (H)
- Standard Control Group (HRZE) (Active Comparator): Standard 6-month regimen. Intensive phase (8 weeks): Rifampicin + Isoniazid + Pyrazinamide + Ethambutol. Consolidation phase (18 weeks): Rifampicin + Isoniazid. Total treatment duration 26 weeks followed by follow-up until week 38.
  Interventions: Drug: Pyrazinamide (PZA); Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Ethambutol (E)

INTERVENTIONS:
Drug: Bedaquiline (B) — Bedaquiline tablets administered orally. Dosing: 400 mg once daily for the first 2 weeks, then 200 mg three times per week for weeks 3-17. Used in both experimental arms (BZMD and BZMH groups) as part of the 4-month short-course regimen for drug-susceptible tuberculosis treatment.
  Other Names: BDQ
  Arms: BZMD Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Delamanid); BZMH Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Isoniazid)
Drug: Moxifloxacin — Moxifloxacin 400 mg tablets administered orally once daily before or after meals throughout the entire treatment period (17 weeks). Used in both experimental arms (BZMD and BZMH groups) as part of the 4-month short-course regimen for drug-susceptible tuberculosis treatment.
  Other Names: Mfx
  Arms: BZMD Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Delamanid); BZMH Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Isoniazid)
Drug: Pyrazinamide (PZA) — Pyrazinamide tablets administered orally once daily in the morning during intensive phase (8 weeks). Dosing by weight: 1000 mg for 40.0-49.9 kg, 1500 mg for 50.0-70.9 kg, 2000 mg for ≥75.0 kg. Used in both experimental arms (BZMD and BZMH groups) and control group as part of tuberculosis treatment regimen.
  Other Names: PZA
Drug: Delamanid (D) — Delamanid tablets administered orally at 100 mg twice daily (total daily dose 200 mg) throughout the entire treatment period (17 weeks). Used only in the BZMD experimental arm as part of the 4-month short-course regimen for drug-susceptible tuberculosis treatment.
  Other Names: Dlm
  Arms: BZMD Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Delamanid)
Drug: Isoniazid (H) — Isoniazid tablets administered orally at 300 mg once daily in the morning throughout the entire treatment period. Used in the BZMH experimental arm (17 weeks) and in the standard control group (26 weeks) as part of tuberculosis treatment regimens.
  Other Names: INH
  Arms: BZMH Group (Bedaquiline + Moxifloxacin + Pyrazinamide + Isoniazid); Standard Control Group (HRZE)
Drug: Rifampicin (R) — Rifampicin tablets administered orally once daily in the morning throughout the entire treatment period (26 weeks). Dosing by weight: 450 mg for 40.0-49.9 kg, 600 mg for 50.0-70.9 kg and ≥75.0 kg. Used only in the standard control group as part of the 6-month standard tuberculosis treatment regimen.
  Other Names: Rif
  Arms: Standard Control Group (HRZE)
Drug: Ethambutol (E) — Ethambutol tablets administered orally during the intensive phase (8 weeks). Dosing by weight: 750 mg for 40.0-49.9 kg, 1000 mg for 50.0-70.9 kg and ≥75.0 kg. Used only in the standard control group as part of the 6-month standard tuberculosis treatment regimen.
  Other Names: Emb
  Arms: Standard Control Group (HRZE)

SUMMARY:
# Brief Summary

This study aims to evaluate the early bactericidal activity (EBA), safety, and tolerability of 4-month short-course regimens containing bedaquiline, moxifloxacin, and pyrazinamide in patients with drug-susceptible tuberculosis. This is a prospective, randomized, controlled, multicenter study planned to enroll 45 rifampicin-susceptible tuberculosis patients, who will be randomized in a 1:1:1 ratio to the BZMD group (bedaquiline + pyrazinamide + moxifloxacin + delamanid), BZMH group (bedaquiline + pyrazinamide + moxifloxacin + isoniazid), and standard control group. Subjects in the test groups will receive 17 weeks (4 months) of group-specific treatment regimens, while subjects in the control group will receive 26 weeks (6 months) of standard HRZE regimen treatment.

The primary endpoint is the change from baseline in log₁₀ colony-forming units (CFU) per milliliter of sputum specimen from Day 0 (pre-dose) to Day 14 of treatment (EBA CFU₀-₁₄), used to evaluate the early bactericidal activity of the drugs. Secondary endpoints include EBA CFU and EBA TTP (time to positive culture) at other time intervals, pharmacokinetic characteristics, sustained microbiological clearance rates, relapse rates, and safety indicators. The study will analyze the daily decline in log₁₀ CFU counts and daily increase in TTP using nonlinear mixed-effects models to reflect the bactericidal activity of the study regimens.

This study will help provide more effective and safer short-course treatment options for Chinese patients with drug-susceptible tuberculosis, thereby improving treatment adherence and treatment success rates, and providing scientific evidence for optimizing short-course treatment regimens for drug-susceptible tuberculosis.

DETAILED DESCRIPTION:
Study Background and Rationale Tuberculosis remains a significant global health challenge, with China ranking among the top three countries with the highest TB burden globally. Current anti-TB treatments for drug-susceptible tuberculosis face major obstacles, primarily poor adherence to long-term (at least 6 months) and complex treatment regimens. Incomplete TB treatment may lead to increased morbidity and mortality, prolonged infectivity, and development of drug resistance.

Recent international studies have demonstrated promising results for shorter treatment regimens. The SimpliciTB study showed that a 4-month short-course regimen containing bedaquiline, moxifloxacin, and pyrazinamide significantly increased 8-week sputum culture clearance rates compared to the standard 6-month regimen. The TRUNCATE-TB study demonstrated that a 2-month regimen containing bedaquiline, isoniazid, and pyrazinamide was non-inferior to standard 6-month treatment. However, bedaquiline-based 4-month short-course regimens have not yet been validated in early-stage studies in the Chinese population.

Study Methodology Treatment Regimens

BZMD Group (Total treatment: 17 weeks):

Intensive phase (8 weeks): Bedaquiline + Pyrazinamide + Moxifloxacin + Delamanid Consolidation phase (9 weeks): Bedaquiline + Moxifloxacin + Delamanid Bedaquiline: 400 mg once daily for 2 weeks, then 200 mg three times weekly for weeks 3-17 Pyrazinamide: Weight-based dosing (1000-2000 mg daily) - intensive phase only Moxifloxacin: 400 mg once daily throughout treatment Delamanid: 100 mg twice daily (200 mg total daily) throughout treatment

BZMH Group (Total treatment: 17 weeks):

Intensive phase (8 weeks): Bedaquiline + Pyrazinamide + Moxifloxacin + Isoniazid Consolidation phase (9 weeks): Bedaquiline + Moxifloxacin + Isoniazid Bedaquiline: Same dosing as BZMD group Pyrazinamide: Weight-based dosing - intensive phase only Moxifloxacin: 400 mg once daily throughout treatment Isoniazid: 300 mg once daily throughout treatment

Standard Control Group (Total treatment: 26 weeks):

Intensive phase (8 weeks): Rifampicin + Isoniazid + Pyrazinamide + Ethambutol Consolidation phase (18 weeks): Rifampicin + Isoniazid

Early Bactericidal Activity Assessment The study employs a rigorous EBA assessment protocol with overnight sputum collections. Subjects must provide at least 10 mL of overnight sputum during each collection cycle. Two pre-treatment overnight sputum specimens are collected on consecutive days before treatment initiation to establish baseline CFU counts. Daily overnight sputum collections continue for the first 14 days of treatment to monitor bactericidal activity.

Pharmacokinetic Substudy A subset of subjects (10-15 per test group) will participate in intensive PK sampling on Day 14, involving 11 blood draws over 24 hours to evaluate steady-state pharmacokinetic characteristics and potential drug-drug interactions between study medications.

Follow-up and Retreatment Criteria All subjects are followed until week 38 post-treatment initiation. For test group subjects who fail to achieve sustained microbiological clearance at end of treatment (week 17) or experience recurrence during follow-up, a standard 6-month HRZE regimen will be re-initiated.

Quality Control Measures

The study implements comprehensive quality assurance including:

* Standardized personnel training for all sites
* Consecutive case enrollment to ensure representativeness
* Dual physician verification of patient information
* Regular monitoring visits by the lead site
* Laboratory quality control with proficiency testing
* Blinded sputum smear rechecking

Statistical Considerations Bactericidal activity will be analyzed using nonlinear mixed-effects models to estimate daily log₁₀ CFU reduction and TTP increases. The study design allows for replacement of subjects who cannot provide adequate sputum specimens to ensure statistical precision. Pharmacokinetic parameters will be compared between test groups using nonparametric methods.

Clinical Significance This study addresses a critical need in tuberculosis treatment by evaluating whether bedaquiline-based short-course regimens can reduce treatment duration from 6 months to 4 months while maintaining efficacy. Successful results could lead to improved treatment adherence, reduced healthcare costs, and decreased risk of drug resistance development. The study specifically focuses on the Chinese population, addressing potential pharmacokinetic and genetic variations that may influence treatment outcomes.

The early bactericidal activity endpoint provides rapid assessment of regimen efficacy, allowing for early identification of promising combinations before larger, longer-term studies. This approach accelerates the development of improved tuberculosis treatment regimens while maintaining rigorous safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤60 years
2. Male or female
3. Body weight 40-90 kg
4. Capable of producing adequate sputum, with collection of at least 10ml overnight sputum
5. Willing to participate in trial treatment and follow-up, with signed informed consent (legal guardian may sign for patients lacking civil capacity)
6. Positive acid-fast bacilli smear microscopy of respiratory specimens (≥1+ according to WHO criteria) and positive rapid amplification test for Mycobacterium tuberculosis in respiratory specimens
7. Rifampicin-susceptible based on molecular drug susceptibility testing or conventional drug susceptibility testing
8. No anti-TB treatment for more than 3 days received within 6 months before the screening period
9. Subjects whose imaging findings meet the diagnostic criteria for TB, as determined by the investigator
10. Women of childbearing potential who have not undergone surgical sterilization must agree to use appropriate contraceptive methods

Exclusion Criteria:

1. Evidence of concurrent extrapulmonary TB
2. Subjects who have participated in other clinical studies within 8 weeks before the screening period
3. Confirmed resistance of mycobacterium tuberculosis isolates to any of the following: Isoniazid, fluoroquinolones, revealed by molecular drug susceptibility testing
4. Known allergy or intolerance to any study drug
5. Patients who cannot receive oral therapy
6. Abnormal liver function (alanine transaminase [ALT], alkaline phosphatase [ALP], or total bilirubin [TBil] exceeding 2 times the upper limit of normal) or known cirrhosis or known alcoholic hepatitis
7. The hematology indicates white blood cells <3.0×10⁹/L, or hemoglobin <80 g/L, or platelets <80×10⁹/L
8. The estimated glomerular filtration rate (eGFR) is less than 60 mL/min/1.73 m²
9. The blood electrolyte test indicates a baseline serum potassium level less than 3.5 mmol/L
10. Subjects who have used drugs known to prolong the QTcF interval for more than 3 days within 30 days before the screening period (including but not limited to amiodarone, bisoprolol, chloroquine, chlorpromazine, cisapride, cyclobenzaprine, clarithromycin, digoxin, dofetilide, domperidone, ertapenem, ibutilide, levomethadone, methadone, pentamidine, quinidine, sotalol, sparfloxacin, thioridazine)
11. Subjects with clinically significant ECG abnormalities as determined by the investigator, including but not limited to: baseline QTcF >450 ms for males or >470 ms for females, presence of second- or third-degree atrioventricular block, QRS duration >120 ms
12. Combined heart failure, coronary artery disease, myocardial infarction, ventricular hypertrophy, clinically significant arrhythmia, poorly controlled hypertension-related cardiovascular disease
13. Patients with known QT prolongation syndrome or a family history thereof
14. Subjects who have used any drug or substance known to be a strong inhibitor of cytochrome P450 enzymes within 30 days before the screening period (including but not limited to ritonavir, ketoconazole, itraconazole, voriconazole, clarithromycin, fluvoxamine, warfarin, rivaroxaban, and other novel oral anticoagulants)
15. Subjects with known bleeding disorders or family history of bleeding disorders
16. Subjects with HIV infection
17. Subjects with known optic neuritis, history of alcoholism, gout, epilepsy, mental illness, porphyria, myasthenia gravis, or malignant tumors
18. Patients with type I or type II diabetes, or HbA1c ≥6.5%, or random blood glucose ≥11.1 mmol/L with typical diabetic symptoms
19. Pregnant or lactating patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Bactericidal Activity CFU 0-14 (EBA CFU₀-₁₄) | Day 0 (baseline) to Day 14 of treatment
  The change from baseline in log10 colony-forming units (CFU) per milliliter of sputum specimen from baseline (Day 0, pre-dose) to Day 14 of treatment. This measures the early bactericidal activity of the drug regimens over the first 14 days of treatment.

SECONDARY OUTCOMES:
Early Bactericidal Activity CFU 0-2 (EBA CFU₀-₂) | Day 0 to Day 2
  The change from baseline in log10 CFU per milliliter of sputum specimen from baseline to Day 2 of treatment.
Early Bactericidal Activity CFU 0-7 (EBA CFU₀-₇) | Day 0 to Day 7
  The change from baseline in log10 CFU per milliliter of sputum specimen from baseline to Day 7 of treatment.
Early Bactericidal Activity TTP 0-14 (EBA TTP₀-₁₄) | Day 0 (baseline) to Day 14 of treatment
  The daily change from baseline in time to positive culture (TTP, in hours) from baseline (Day 0, pre-dose) to Day 14 of treatment. This measures the early bactericidal activity by evaluating the extension in time required for bacterial culture to become positive.
Sustained Microbiological Clearance Rate | Week 17 (end of treatment)
  The sustained microbiological clearance rate at the end of 17 weeks of treatment in the test groups and control group. Defined as at least two consecutive negative culture results from respiratory specimens after baseline, with an interval of ≥14 days between specimen collection dates.
Safety - Grade 3 or Higher Adverse Events | From enrollment through study completion, up to 52 weeks
  Occurrence of Grade 3 or above adverse events according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) criteria during the study period.

OTHER OUTCOMES:
Early Bactericidal Activity CFU 7-14 (EBA CFU₇-₁₄) | Day 7 to Day 14 of treatment
  The change from baseline in log10 colony-forming units (CFU) per milliliter of sputum specimen from Day 7 to Day 14 of treatment. This measures the bactericidal activity during the second week of treatment.
Early Bactericidal Activity TTP 0-2 (EBA TTP₀-₂) | Day 0 (baseline) to Day 2 of treatment
  The daily change from baseline in time to positive culture (TTP, in hours) from baseline (Day 0, pre-dose) to Day 2 of treatment. This measures the very early bactericidal activity within the first 2 days of treatment.
Early Bactericidal Activity TTP 0-7 (EBA TTP₀-₇) | Day 0 (baseline) to Day 7 of treatment
  The daily change from baseline in time to positive culture (TTP, in hours) from baseline (Day 0, pre-dose) to Day 7 of treatment. This measures the early bactericidal activity during the first week of treatment.
Early Bactericidal Activity TTP 7-14 (EBA TTP₇-₁₄) | Day 7 to Day 14 of treatment
  The daily change from baseline in time to positive culture (TTP, in hours) from Day 7 to Day 14 of treatment. This measures the bactericidal activity during the second week of treatment by evaluating changes in time to culture positivity.
Relapse Rate | Up to Week 52 (end of follow-up phase)
  The relapse rate in the test groups and control group at the end of the follow-up phase. Relapse is defined as subjects who had previously received anti-TB treatment in the regimen, were judged as cured or completed treatment at the end of treatment, and are now diagnosed with tuberculosis (whether relapse or reinfection).
AUC₀-₂₄ of Anti-TB Drugs | Day 14 (24-hour intensive sampling)
  Area under the concentration-time curve from 0 to 24 hours (AUC₀-₂₄) at steady-state for Bedaquiline, Moxifloxacin, Pyrazinamide, Delamanid, and Isoniazid.
Cmax of Anti-TB Drugs | Day 14 (24-hour intensive sampling)
  Maximum plasma concentration at steady-state (Cₘₐₓ,ₛₛ) for Bedaquiline, Moxifloxacin, Pyrazinamide, Delamanid, and Isoniazid.
Adverse Drug Reactions | From enrollment through study completion, up to 52 weeks
  Occurrence of adverse drug reactions (ADRs) that are determined to be related to the study medications. ADRs are defined as adverse events with evidence of reasonable temporal relationship with study drug use and more likely attributable to the study drug than to other causes.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this study will be shared, including:
  1. Efficacy data: Early bactericidal activity measurements (CFU counts, time to positive culture), sustained microbiological clearance rates, and relapse rates
  2. Safety data: Adverse events, serious adverse events, laboratory values, and vital signs
  3. Pharmacokinetic data: Drug concentration measurements and calculated PK parameters for participants who consented to PK sampling
  4. Demographic and baseline characteristics: Age, sex, body weight, baseline disease characteristics, and medical history
  5. Treatment data: Drug dosing, treatment duration, adherence, and treatment modifications Data will be shared after de-identification and removal of all direct and indirect identifiers. The study protocol, statistical analysis plan, informed consent form, and clinical study report will also be made available.

REFERENCES:
- [Background] Paton NI, Cousins C, Suresh C, Burhan E, Chew KL, Dalay VB, Lu Q, Kusmiati T, Balanag VM, Lee SL, Ruslami R, Pokharkar Y, Djaharuddin I, Sugiri JJR, Veto RS, Sekaggya-Wiltshire C, Avihingsanon A, Sarin R, Papineni P, Nunn AJ, Crook AM; TRUNCATE-TB Trial Team. Treatment Strategy for Rifampin-Susceptible Tuberculosis. N Engl J Med. 2023 Mar 9;388(10):873-887. doi: 10.1056/NEJMoa2212537. Epub 2023 Feb 20. PMID 36808186
- [Background] Cevik M, Thompson LC, Upton C, Rolla VC, Malahleha M, Mmbaga B, Ngubane N, Abu Bakar Z, Rassool M, Variava E, Dawson R, Staples S, Lalloo U, Louw C, Conradie F, Eristavi M, Samoilova A, Skornyakov SN, Ntinginya NE, Haraka F, Praygod G, Mayanja-Kizza H, Caoili J, Balanag V, Dalcolmo MP, McHugh T, Hunt R, Solanki P, Bateson A, Crook AM, Fabiane S, Timm J, Sun E, Spigelman M, Sloan DJ, Gillespie SH; SimpliciTB Consortium. Bedaquiline-pretomanid-moxifloxacin-pyrazinamide for drug-sensitive and drug-resistant pulmonary tuberculosis treatment: a phase 2c, open-label, multicentre, partially randomised controlled trial. Lancet Infect Dis. 2024 Sep;24(9):1003-1014. doi: 10.1016/S1473-3099(24)00223-8. Epub 2024 May 17. PMID 38768617
- [Background] Tasneen R, Garcia A, Converse PJ, Zimmerman MD, Dartois V, Kurbatova E, Vernon AA, Carr W, Stout JE, Dooley KE, Nuermberger EL. Novel Regimens of Bedaquiline-Pyrazinamide Combined with Moxifloxacin, Rifabutin, Delamanid and/or OPC-167832 in Murine Tuberculosis Models. Antimicrob Agents Chemother. 2022 Apr 19;66(4):e0239821. doi: 10.1128/aac.02398-21. Epub 2022 Mar 22. PMID 35315690
- See also: World Health Organization Global Tuberculosis Report 2024 providing epidemiological background and current treatment recommendations for drug-susceptible tuberculosis. — https://iris.who.int/handle/10665/379339
- See also: WHO consolidated guidelines on drug-susceptible tuberculosis treatment providing evidence-based recommendations for standard treatment regimens and management approaches that inform the study design and comparator arm selection. — https://www.who.int/publications/i/item/9789241550529